CLINICAL TRIAL: NCT04874038
Title: Prevention of Persistent Pain With LidocAine iNfusions in Breast Cancer Surgery (PLAN)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-5021
Record Dates: First submitted 2021-04-20; First posted 2021-05-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Post-mastectomy Pain Syndrome; Breast Cancer; Pain, Postoperative; Pain, Chronic
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Chronic Pain | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intraoperative intravenous lidocaine/placebo infusion
  Interventions: Drug: Lidocaine 20mg/ml
- Control (Placebo Comparator): Intraoperative intravenous lidocaine/placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine 20mg/ml — Patients in the intervention group will receive an IV lidocaine infusion using a dosage regimen of 1.5 mg/kg bolus of a 2% lidocaine solution with induction of general anesthesia followed by a 2.0 mg/kg/hour infusion until the end of surgery (and up to 30 minutes into recovery room).
  Other Names: Lidocaine 2%
  Arms: Intervention
Drug: Placebo — Patients in the control group will receive a placebo bolus and infusion with normal saline (0.9% sodium chloride solution) until the end of surgery (and up to 30 minutes into recovery room).
  Other Names: 0.9% sodium chloride solution
  Arms: Control

SUMMARY:
Phase III, international multicentre, parallel group, blinded, 1:1 randomized controlled trial to determine the effect of an intraoperative intravenous lidocaine infusion on reducing the development of persistent pain 3-months after breast cancer surgery.

DETAILED DESCRIPTION:
PLAN is a multicentre, parallel-group, blinded, randomized controlled trial of 1,602 patients undergoing breast cancer surgery. Consented eligible patients will be randomized to receive an intravenous lidocaine: 1.5 mg/kg bolus with induction of general anesthesia followed by a 2.0 mg/kg/hour infusion until the end of surgery (and up to 30 minutes into recovery room). Patients in the control group will receive a placebo bolus and infusion with normal saline (0.9% sodium chloride solution). Study medications will be prepared in blinded 50 mL syringes and labelled as per Regulatory requirements. Patients will follow up on the first 3 days after surgery, and at 3 and 12-months postoperatively to report on pain, analgesic consumption, functional, mood, and quality of life outcomes

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Undergoing a unilateral or bilateral lumpectomy or mastectomy, inclusive of all pathologies, including prophylactic surgery (e.g., family history or BRCA gene mutation)

Exclusion Criteria:

1. Previous breast surgery within 6 months of index surgery
2. Undergoing any autologous flap procedure during index surgery
3. Presence known chronic pain disorder involving surgical site or ipsilateral chest wall, shoulder, or arm during the 3-months prior to index surgery
4. Documented hypersensitivity or allergy to lidocaine
5. Surgery not planned to be performed under general anesthesia and/or planned use of regional or neuraxial anesthetic techniques before surgery (i.e., epidural, paravertebral, serratus plane block, pectoralis or modified pectoralis block)
6. History of ventricular tachycardia, ventricular fibrillation, or atrioventricular block without a pacemaker
7. Known cirrhotic liver disease
8. Pregnant
9. Unlikely to comply with follow-up (e.g. no fixed address, language difficulties that would impede valid completion of questionnaires, plans to move out of town)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1602 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Development of persistent pain 3-months after breast cancer surgery | 3- months
  Persistent pain at 3-months

SECONDARY OUTCOMES:
Pain intensities | 3 and 12 months
  Pain intensities measured on the Numeric Rating Scale (NSR) at rest and movement.
Opioid consumption | 3 and 12 months
  Morphine-equivalent opioid consumption
Moderate-to-severe persistent pain | 3 and 12 months
  Defined as persistent pain with an NRS pain score of ≥4 at rest 24-hours
Persistent neuropathic pain | 3 and 12 months
  Measured using the Douleur Neuropathique 4-symptoms interview
Sensory and affective qualities of pain | 3 and 12 months
  Quality of pain is reported using the Short Form McGill Pain Questionnaire
Emotional functioning | 3 and 12 months
  Emotional functioning is reported using the Profile of Mood States (POMS)
Physical functioning | 3 and 12 months
  Physical functioning measured by the interference scale of the Brief Pain Inventory-Short Form.
Health-related quality of life quality of life | 3 and 12 months
  Health-related quality of life will be assessed using EQ-5D-5L
Cancer Recurrence | 3 and 12 months
  Cancer recurrence will be assessed as a secondary outcome
Adverse events | 3 and 12 months
  Adverse Events will be monitored as a secondary safety outcome
Cost Effectiveness | 3 months
  Healthcare Costs associated with the burden of chronic post-surgical pain will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: James Khan, MD, Principal Investigator — University Health Network, Toronto; PJ Devereaux, MD.PhD, Principal Investigator — Population Health Research Institute; Ian Gilron, MD, Principal Investigator — Kingston Health Sciences Centre
Locations (17):
- Canada (15):
  - Foothills Medical Centre, Calgary, Alberta
  - Sturgeon Community Hospital, Edmonton, Alberta
  - Eastern Health- Health Sciences Centre, St. John's, Newfoundland and Labrador
  - IWK, Halifax, Nova Scotia
  - Juravinski Hospital, Hamilton, Ontario
  - North York General Hospital, North York, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- B.P. Koirala Institute of Health Sciences, Dharān, Nepal
- Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan JS, Gilron I, Devereaux PJ, Clarke H, Ayach N, Tomlinson G, Quan ML, Ladha KS, Choi S, Munro A, Brull R, Lim DW, Avramescu S, Richebe P, Hodgson N, Paul J, McIsaac DI, Derzi S, Zbitnew GL, Easson AM, Siddiqui NT, Miles SJ, Karkouti K; PLAN Trial Investigators. Prevention of persistent pain with lidocaine infusions in breast cancer surgery (PLAN): study protocol for a multicenter randomized controlled trial. Trials. 2024 May 22;25(1):337. doi: 10.1186/s13063-024-08151-4. PMID 38773653